CLINICAL TRIAL: NCT05603572
Title: A Multi-center, Open-label, Phase 1/2a Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of KAT-101 in Subjects With HCC
Brief Title: KAT-101 in Subjects With Hepatocellular Carcinoma (HCC)
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enrollment paused
Sponsor: Primocure Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NLP-KAT-101
Record Dates: First submitted 2022-10-23; First posted 2022-11-02 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Hepatocellular Carcinoma; Fibrolamellar Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrolamellar hepatocellular carcinoma

STUDY DESIGN:
Intervention Model Description: 1. Oral administration (KAT-101)
  2. IT administration (KAT-201)
  3. Oral administration (KAT-101) + IT administration (KAT-201)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Oral experimental arm (Experimental): Oral administration (KAT-101) taken once per day for 4 consecutive days out of 7 (4 days on / 3 days off weekly). Each cycle is 28 days. Treatment will continue for up to 12 cycles until progressive disease (PD), unacceptable toxicity, or any reason for discontinuing its administration, whichever occurs first.
  Interventions: Drug: KAT-101
- IT experimental arm (Experimental): IT administration (KAT-201) will be injected via percutaneous IT injection with ultrasound and/or computed tomography (CT) guidance once a week (on Day 1 weekly). Each cycle is 28 days. Treatment will continue for up to 2 cycles until PD, unacceptable toxicity, or any reason for discontinuing its administration, whichever occurs first.
  Interventions: Drug: KAT-201
- Oral + IT experimental arm (Experimental): Once optimal oral and IT dose are determined, oral + IT will be administered as follows: oral administration (KAT-101) will be taken once per day for 4 consecutive days out of 7 (4 days on / 3 days off weekly). Treatment will continue for up to 12 cycles (each cycle 28 days). IT administration (KAT-201) will be injected via percutaneous IT injection with ultrasound and/or CT guidance once a week (on Day 1 weekly). Treatment will continue for up to 2 cycles (each cycle 28 days) until PD, unacceptable toxicity, or any reason for discontinuing its administration, whichever occurs first.
  Interventions: Drug: KAT-101; Drug: KAT-201

INTERVENTIONS:
Drug: KAT-101 — oral dosage form
  Arms: Oral + IT experimental arm; Oral experimental arm
Drug: KAT-201 — IT dosage form
  Arms: IT experimental arm; Oral + IT experimental arm

SUMMARY:
NLP-KAT-101 is a Phase 1/2a dose escalation and expansion study to investigate the safety, tolerability, PK, and preliminary efficacy of oral + intratumoral (IT) KAT in subjects with HCC.

DETAILED DESCRIPTION:
Phase 1 will identify the optimal dose for oral alone, IT alone and the recommended Phase 2 dose (RP2D) dose for oral + IT together. Once the RP2D is identified, additional subjects will be enrolled into Phase 2a (dose-expansion) to further investigate the efficacy and safety of oral + IT KAT at the RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HCC not amenable to surgical resection or curative-intent locoregional ablative treatments and who are not eligible for liver transplantation.
* Systemic treatment-naive for unresectable locally advanced or metastatic HCC. In addition, have progressed on, refused or were intolerant to sorafenib, lenvatinib, or atezolizumab in combination with bevacizumab. A maximum of 2 prior lines of systemic therapy (including chemotherapy or targeted therapy, not including locoregional therapy) will be allowed.
* At least one measurable lesion based on RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate organ function

Exclusion Criteria:

* Prior to the first administration of the study treatment:

  1. Major surgery within 28 days
  2. Radiotherapy within 14 days including palliative radiation
  3. Use of steroids (except for topical agents) within 14 days
  4. Chemotherapy within 3 weeks (6 weeks for nitrosourea compounds)
  5. Prior treatment with biologic agents, including hormone therapy, within the last 3 weeks, or at least 5 half-lives, whichever is shorter
  6. Tumor infiltration in the portal vein, hepatic veins or inferior vena cava that completely blocks circulation in liver
  7. Treatment with another investigational product within 4 weeks prior to screening or for which 5 half-lives have not elapsed, whichever is longer
  8. Uncontrolled central nervous system (CNS) metastasis
* Any clinically significant abnormal intestinal findings that may interfere with the investigational product
* Severe cardiac disorders or subjects with comorbidities of other serious internal disorders on investigator's judgment
* QTcF > 450 msec or congenital long QT syndrome
* Suspected serious infectious diseases, intestinal paralysis, bowel obstruction, interstitial pneumonia, or pulmonary fibrosis
* Serious underlying medical or psychiatric condition, dementia or altered mental status that would impair the ability to understand informed consent, contraindicate participation in the study or confound the results of the study
* Known human immunodeficiency virus (HIV) infection or chronic or active hepatitis B virus (HBV) hepatitis C virus (HCV). Subjects with HCV who have a documented cure (undetectable HCV ribonucleic acid (RNA) 24 weeks after the end of treatment) may be enrolled.
* Severe physical or mental trauma that results from injury or a wound(s).
* Any condition or non-removable device contraindicated for MRI examination
* Pregnant women or nursing mothers.
* Women of childbearing potential (WOCBP) who are unwilling to use a medically acceptable method of birth control during the study until 185 days after the last dose of study treatment
* Men with partners of childbearing potential who are unwilling to use condoms in combination with a second medically acceptable method of contraception during the study until 95 days after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
To determine the Recommended Phase 2 Dose (RP2D) for oral + IT administration | 24 months
  RP2D is defined as the dose at which dose escalation (oral + IT) ceases

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of KAT (oral, IT, and oral + IT) in subjects with HCC | 54 months
  Measured as the number of AEs per CTCAE and changes in laboratory values compared to baseline.
To evaluate the preliminary anti-tumor activity of KAT for oral + IT administration | 54 months
  Overall response rate (ORR) is defined as the proportion of subjects with a best overall response (BOR) by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) and/or mRECIST; disease control rate (DCR), defined as the proportion of subjects with a BOR of CR, PR, or stable disease (SD); duration of response (DOR), defined as the length of time from the time of response (CR or PR) to the time of PD or death; progression-free survival (PFS), defined as the time from the date of treatment initiation to PD or death; overall survival (OS), defined as the length of time from the date of treatment initiation to death from any cause.
To assess maximum concentration (Cmax) of KAT (oral and oral + IT) | 54 months
  Blood samples will be drawn to determine Cmax of KAT
To assess median time to the maximum drug concentration (Tmax) of KAT (oral and oral + IT) | 54 months
  Blood samples will be drawn to determine Tmax of KAT
To assess half lives (T1/2) of KAT (oral and oral + IT) | 54 months
  Blood samples will be drawn to determine T1/2 of KAT
To assess area under the curve (AUC) of KAT (oral and oral + IT) | 54 months
  Blood samples will be drawn to determine AUC of KAT

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Kyungpook National University Hospital, Daegu
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No